COMIRB
APPROVED
For Use

Study Title: Engaging Practices and Communities in the Development of Interventions to Promote 03-Jul-2021 HPV Vaccine Uptake

Principal Investigator: Sean O'Leary, MD, MPH

**COMIRB No: 18-0338** 

Version Date: June 11, 2021

You are being asked to be in this research study because you participated in the design process or dissemination of community vaccine education materials.

If you join the study, you will participate in an interview that lasts up to 30-45 minutes. You will receive a compensation in the form of a \$25 electronic gift card for your time.

This study is designed to learn more about the impacts of BCT developed materials on HPV vaccine uptake.

Possible discomforts or risks include a small chance that people will feel uncomfortable answering questions about vaccines. There may be risks the researchers have not thought of. This study is not designed to benefit you directly.

Every effort will be made to protect your privacy and confidentiality by storing and analyzing all demographic information, audio files, and interview transcripts on encrypted computers inside the University firewall

This research is being paid for by the National Institutes of Health.

You have a choice about being in this study. You do not have to be in this study if you do not want to be

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

If you have questions, you can call Dr. Sean O'Leary at 303-724-1582. You can call and ask questions at any time.

You may have questions about your rights as someone in this study. If you have questions, you can call COMIRB (the responsible Institutional Review Board) at (303) 724-1055.

By completing this survey, you are agreeing to participate in this research study.